CLINICAL TRIAL: NCT00517608
Title: Monopolar Scissors vs Bipolar Vessel Sealer vs Ultrasonic Shears: A Prospective Randomized Study in Laparoscopic Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-2005
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Colorectal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Laparoscopic colectomy

SUMMARY:
Monopolar electro surgery scissors (MES), electro thermal bipolar vessel sealer (BVS) and ultrasonically coagulating shears (UCS) are all applied in laparoscopic colorectal surgery. We aimed to compare the different devices with regard to dissection time, blood loss, technical aspects and costs.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria: All patients undergoing laparoscopic left-sided colorectal resection.

Exclusion criteria: < 18 years no informed consent restricted communication abilities (language, mental illness)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Dissection time

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Hubner M, Demartines N, Muller S, Dindo D, Clavien PA, Hahnloser D. Prospective randomized study of monopolar scissors, bipolar vessel sealer and ultrasonic shears in laparoscopic colorectal surgery. Br J Surg. 2008 Sep;95(9):1098-104. doi: 10.1002/bjs.6321. PMID 18690630